CLINICAL TRIAL: NCT03056482
Title: Haloperidol Versus Ondansetron for Cannabis Hyperemesis Syndrome (HaVOC): A Randomized Controlled Trial
Brief Title: Haloperidol Versus Ondansetron for Cannabis Hyperemesis Syndrome (HaVOC)
Acronym: HaVOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Marco L.A. Sivilotti (Other)
Responsible Party: Sponsor-Investigator, Dr. Marco L.A. Sivilotti, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMED-251-17
Record Dates: First submitted 2017-01-23; First posted 2017-02-17 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cannabis Use Disorder
Keywords: cannabis; haloperidol; ondansetron; hyperemesis; cyclic vomiting syndrome
MeSH Terms: conditions — Marijuana Abuse; Hyperemesis Gravidarum; Familial cyclic vomiting syndrome | interventions — Ondansetron; Haloperidol

STUDY DESIGN:
Intervention Model Description: This is a double-blinded, randomized, cross-over clinical trial that will allocate subjects in a 1:1:1 fashion into one of three treatment groups: high- or low-dose haloperidol, or ondansetron, with a minimum 7-day washout period between treatments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be allocated to an intervention via a sealed, opaque envelope system to be opened by an unblinded nurse not otherwise involved in patient care or research procedures will prepare the intervention. The Attending physician, Research personnel and Investigator(s) will all remain blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ondansetron 8mg (Active Comparator): 8mg Ondansetron prepared in a 100mL normal saline mini-bag
  Interventions: Drug: Ondansetron 8mg
- Haloperidol 0.05mg/kg (Experimental): 0.05mg/kg of Haloperidol prepared in a 100mL normal saline mini-bag
  Interventions: Drug: Haloperidol 0.05mg/kg
- Haloperidol 0.1mg/kg (Experimental): 0.1mg/kg of Haloperidol prepared in a 100mL normal saline mini-bag
  Interventions: Drug: Haloperidol 0.1mg/kg

INTERVENTIONS:
Drug: Ondansetron 8mg — Ondansetron 8 MG prepared in a 100 mL normal saline min-bag
  Other Names: Zofran
  Arms: Ondansetron 8mg
Drug: Haloperidol 0.05mg/kg — Haloperidol 0.05 mg/kg prepared in a 100 mL normal saline min-bag
  Other Names: Haldol
  Arms: Haloperidol 0.05mg/kg
Drug: Haloperidol 0.1mg/kg — Haloperidol 0.1 mg/kg prepared in a 100 mL normal saline min-bag
  Other Names: Haldol
  Arms: Haloperidol 0.1mg/kg

SUMMARY:
Cannabis Hyperemesis Syndrome (CHS) has become a well-documented syndrome since 2004 and is expected to increase in prevalence with continuing liberalization of marijuana and recognition of the disease. Regardless of whether the association with heavy cannabis use is recognized, there is well-documented resistance to traditional anti-emetic treatment. Given promising reports of the use of intravenous haloperidol, a randomized controlled trial comparing it to the commonly administered anti-emetic ondansetron will contribute to the management of CHS

DETAILED DESCRIPTION:
This is a double-blinded, randomized, cross-over clinical trial that will enroll approximately 80 subjects from at least four different research sites. Patients who have been diagnosed with CHS and enrolled in our study will act as their own controls upon their return to the ED for a subsequent bout of CHS for up to 3 visits per subject. Each patient will be allocated in a 1:1:1 fashion into one of three treatment groups: high- or low-dose haloperidol, or ondansetron, with a minimum 7-day washout period between treatments. As CHS tends to be a recurrent syndrome (presumably given the continued use of cannabis despite recommendations to taper and abstain), it is expected that most subjects will return at least once again, and a substantial subset of the study population will complete all three treatment visits during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Self-report of ≥3 episodes of emesis occurring in a cyclic pattern for greater than 1 month in the preceding 2 years
3. Current episode >2 hours of emesis
4. At least one episode of emesis/forceful retching witnessed (including products of emesis at bedside) or heard by an independent observer (healthcare provider or family/friend) in the emergency department
5. Self-reported frequent (near daily to daily x at least 6 months) use of cannabis by inhalation.
6. Working diagnosis of cannabis hyperemesis syndrome in the opinion of the treating emergency physician

Exclusion Criteria:

1. Chronic, daily use of opioid equivalent to ≥10mg morphine/day
2. Inability to comprehend study consent or instructions
3. Unreliable follow-up/unlikely to return for cross-over
4. Administration of an intravenous antiemetic, anticholinergic or antipsychotic (other than up to 100mg dimenhydrinate) in the previous 24 hours
5. Allergy or intolerance to haloperidol or ondansetron
6. Pregnancy
7. Any other medical or psychiatric condition that in the opinion of the enrolling physician would interfere with participation in the trial
8. Current active participation in an investigational drug trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-21 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Change in pain and nausea | 2 hours
  Difference between arithmetic mean of Pain Score and Nausea Score (each on a 10-cm VAS) at 2 hours versus at baseline

SECONDARY OUTCOMES:
Change in pain | 1, 2, 24 and 48 hours
  Changes in abdominal pain score at 1, 2, 24 and 48 hours vs. baseline
Change in nausea | 1, 2, 24 and 48 hours
  Changes in nausea score at 1, 2, 24 and 48 hours vs. baseline
Treatment success | 2, 24 and 48 hours
  Treatment success = both abdominal pain and nausea score < 2 at 2, 24 and 48 hours
Oral intake | 2 hours
  Cumulative oral intake from t=0 to 2 hours (in mL)
Emesis volume | 2 hours
  Cumulative emesis from t=0 to 2 hours (in mL)
Urine output | 2 hours
  Cumulative urine output (in mL)
Discharge ready at 2 hours | 2 hours
  Deemed discharge-ready at 2 hours in the opinion of the treating physician
Rescue anti-emetics in ED | at discharge from Emergency Department or 12 hours whichever comes first
  Given rescue anti-emetics prior to discharge
Time to discharge from ED | at discharge from Emergency Department or 12 hours whichever comes first
  Time interval to discharge-ready from t=0 (min)
Subject preferred arm | 2 hours
  Subject preference of high- vs low-dose haloperidol, and of haloperidol vs ondansetron (-10, 10)
Return to ED | 7 days
  Unscheduled return visits to ED within 7 days (count)
ED consult | From time of study intervention until admitting service consulted or subject discharged from Emergency Department, whichever comes first, assessed up to 48 hours
  Consulted to admitting service
Prolonged ED Length of stay | at discharge from Emergency Department or 12 hours whichever comes first
  Outcome 10 "Time to Discharge from ED" > 12 hours (binary yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Marco LA Sivilotti, MD, MSc, Principal Investigator — Dept. of Emergency Medicine, Queen's University
Locations (3):
- Canada (3):
  - Hotel Dieu Hospital, Kingston, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Queen's University, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruberto AJ, Sivilotti MLA, Forrester S, Hall AK, Crawford FM, Day AG. Intravenous Haloperidol Versus Ondansetron for Cannabis Hyperemesis Syndrome (HaVOC): A Randomized, Controlled Trial. Ann Emerg Med. 2021 Jun;77(6):613-619. doi: 10.1016/j.annemergmed.2020.08.021. Epub 2020 Nov 5. PMID 33160719